CLINICAL TRIAL: NCT06921733
Title: Non-invasive Evaluation of Kidneys in Patient With Congenital Anomalies of the Kidney and Urinary Tract (CAKUT) Using Ultrasound Localization Microscopy
Brief Title: Ultrasound Localization Microscopy in Patient With Congenital Anomalies of the Kidney and Urinary Tract (CAKUT)
Acronym: Search_CAKUT
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, PD Dr. med. Dr. rer. biol. hum. Ferdinand Knieling, University Hospital Erlangen
Other Study IDs: Search_CAKUT_ULM
Record Dates: First submitted 2024-10-21; First posted 2025-04-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Congenital Anomalies of Kidney and Urinary Tract; Lower Urinary Tract Obstruction, Congenital; Ureteropelvic Junction Obstruction; Hydronephrosis Congenital
MeSH Terms: conditions — Cakut; Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with congenital anomalies of the kidney and urinary tract (CAKUT) with indication for MAG3: Included will be children under the age of 6 with congenital anomalies of the kidney and urinary tract (CAKUT)that get an indication for a MAG3 scintigraphy. They will be monitored with CEUS/ULM after the MAG3 scintigraphy.
  Interventions: Device: Contrast enhanced ultrasound imaging (CEUS) and post processing with ULM

INTERVENTIONS:
Device: Contrast enhanced ultrasound imaging (CEUS) and post processing with ULM — CEUS is a contrast based ultrasound technique and ULM (Ultrasound Localization Microscopy) is a post-processing bioinformatical method to quantify microvascular architecture and perfusion dynamics.

SUMMARY:
This clinical study aims to non-invasively visualize perfusion and microvascularization, as well as individual glomeruli, using Ultrasound Localization Microscopy (ULM) and CEUS in patients with congenital anomalies of the kidney and urinary tract (CAKUT).

DETAILED DESCRIPTION:
Congenital anomalies of the kidney and urinary tract (CAKUT) affect 0.5% of newborns and account for 20% of all congenital malformations. These conditions are associated with chronic kidney failure, a need for dialysis, and significantly increased mortality (30 times higher than healthy peers) and morbidity. Patients with CAKUT face substantial health and socioeconomic burdens due to lifelong therapy requirements. In Europe, CAKUT is the leading cause of dialysis-dependent chronic kidney failure.

All CAKUT disorders arise in utero, interfering with kidney development and leading to reduced nephron formation. Many congenital kidney anomalies are diagnosed via prenatal ultrasound. These anomalies include ureteropelvic junction obstruction, often presenting as unilateral hydronephrosis, and posterior urethral valves, which can be associated with megacystis and bilateral hydronephrosis. The resulting urinary obstruction can cause pressure damage to kidney tissue during fetal development, further reducing functional nephron mass. Postnatally, ongoing pressure damage can lead to renal remodeling. The decreased nephron mass and remodeling increase the long-term risk of kidney insufficiency, which is currently assessed only by serum creatinine levels-these are delayed and less sensitive in infants and young children. Reliable biomarkers for reduced nephron mass or renal remodeling to predict chronic kidney injury risk in CAKUT patients are currently lacking. Currently, the actual pressure impact of sonographically detectable urinary obstruction can only be assessed through urine flow patterns using MAG-3 scintigraphy. However, this method is dependent on kidney function, which can affect the uptake and excretion of the radiopharmaceutical and subsequently influence the evaluation of results.

The intravenous use of ultrasound contrast enhancers as an aid opens up the possibility of recording the tissue perfusion of the kidneys, including the smallest vessels, independent of the kidney function. This could provide significantly more information compared to conventional methods and expand our knowledge of the pathophysiology and individual status of tissue perfusion in patients.

In this clinical study, the new CEUS measurement and imaging technique will be used after the kidney scintigraphy. A contrast agent (SonoVue®) will be administered during the routine ultrasound examination and improved tissue visualization will be achieved. The aim is to gain new insights into kidney perfusion as part of the treatment and to better assess the extent of organ damage in the individual patient through more specific vascular imaging. Finally, the aim is to compare diagnostic and prognostic methods with the currently recommended measures. The CEUS is to be examined as a possible diagnostic imaging tool and possibly a supplement to existing diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

Minimum Age 1 Month Maximum Age 6 Years Indication for MAG3 Scintigraphy of the Kidney Congenital Anomalies of the Kidney and Urinary Tract Obstruction Diagnosis Availability of the qualified examiner Consent of the parents/legal guardians

Exclusion Criteria:

Lack of consent of at least one parent

Ages: 0 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One study population. Anticipated approx. n=20 children with above mentioned inclusion criteria with congenital anomalies of the kidney and urinary tract and inclusion criteria for MAG3 scintigraphy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
CEUS Measurement1 | Baseline and follow up (1-31 days after routine surgery if indicated)
  PE (Peak-Enhancement)
CEUS Time intensity curves | Baseline and follow up (1-31 days after routine surgery if indicated)
  All CEUS outcomes will be generated in order to achieve time intensity curves in contrast enhanced ultrasound analysis
CEUS Measurement2 | Baseline and follow up (1-31 days after routine surgery if indicated)
  WiAUC (Wash-in Area Under the Curve (AUC(TI: TTP)))
CEUS Measurement4 | Baseline and follow up (1-31 days after routine surgery if indicated)
  RT (Rise Time)
CEUS Measurement5 | Baseline and follow up (1-31 days after routine surgery if indicated)
  mTT (mean Transit Time local) (mTT-TI))
CEUS Measurement6 | Baseline and follow up (1-31 days after routine surgery if indicated)
  TTP (Time to Peak)
CEUS Measurement7 | Baseline and follow up (1-31 days after routine surgery if indicated)
  WiR (Wash-in-Rate )
CEUS Measurement8 | Baseline and follow up (1-31 days after routine surgery if indicated)
  WiPI (Wash-in Perfusion Index (WiAUC/RT))
CEUS Measurement9 | Baseline and follow up (1-31 days after routine surgery if indicated)
  WoAUC (Wash-out AUC (AUC(TTP:TO)))
CEUS Measurement10 | Baseline and follow up (1-31 days after routine surgery if indicated)
  WiWoAUC (Wash-in- und Wash-out-AUC (WiAUC+WoAUC))
CEUS Measurement11 | Baseline and follow up (1-31 days after routine surgery if indicated)
  FT (Fall Time - (TO-TTP))
CEUS Measurement12 | Baseline and follow up (1-31 days after routine surgery if indicated)
  WOR (Wash-out-Rate) QOF (Quality Of Fit between the echo-power signal and f(t)
CEUS Measurement13 | Baseline and follow up (1-31 days after routine surgery if indicated)
  QOF (Quality Of Fit between the echo-power signal and f(t)
Visualization and quantification of kidney perfusion with CEUS | Baseline and follow up (1-31 days after routine surgery if indicated)
  CEUS imaging for kidney perfusion in CAKUT
Visualization and quantification of kidney mikrovaskularisation with ULM | Baseline and follow up (1-31 days after routine surgery if indicated)
  ULM imaging for kidney perfusion and mikrovaskularisation in CAKUT
Visualization and quantification of glomeruli in the kidney with ULM | Baseline and follow up (1-31 days after routine surgery if indicated)
  ULM imaging for glomeruli in the kidney

SECONDARY OUTCOMES:
ULM and Ultrasound | Baseline and follow up (1-31 days after routine surgery if indicated)
  Correlation of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) with sonographic parameters (including Resistance Index (RI), flow velocity).
ULM and CEUS | Baseline and follow up (1-31 days after routine surgery if indicated)
  Correlation of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) with parameters of contrast-enhanced ultrasound (CEUS).
ULM and Biopsy | Baseline and follow up (1-31 days after routine surgery if indicated)
  Correlation of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (including the number of segmented glomeruli) with histological parameters.
ULM on affected and unaffected kidney | Baseline and follow up (1-31 days after routine surgery if indicated)
  Comparison of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) between the affected and unaffected kidney in the same patient.
ULM and Scintigraphy | Baseline and follow up (1-31 days after routine surgery if indicated)
  Correlation of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) with parameters from renal scintigraphy (e.g., perfusion parameters).
Pressure changes with CEUS | Baseline and follow up (1-31 days after routine surgery if indicated)
  Visualization of pressure changes in the kidney using the vascular architecture visualized by CEUS and parameters of quantified microvascular perfusion dynamics.
Pressure changes with ULM | Baseline and follow up (1-31 days after routine surgery if indicated)
  Visualization of pressure changes in the kidney using the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics.
Comparison of the kidney before and after intervention with ULM | Baseline and follow up (1-31 days after routine surgery if indicated)
  Comparison of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) before and after intervention
ULM on different diagnoses | Baseline and follow up (1-31 days after routine surgery if indicated)
  Comparison of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) between different diagnoses.
ULM on clinical outcomes | Baseline and follow up (1-31 days after routine surgery if indicated)
  Correlation and comparison of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) with clinical criteria and clinical outcomes (surgical success).
Correlation between ULM and laboratory parameters | Baseline and follow up (1-31 days after routine surgery if indicated)
  Correlation of the vascular architecture visualized by ULM and parameters of quantified microvascular perfusion dynamics of the kidney (e.g., number of segmented glomeruli) with laboratory parameters (including kidney function parameters, inflammatory markers, and immunological parameters).
Assessment of renal function GFR | Baseline and follow up (1-31 days after routine surgery if indicated)
  GFR (ml/min/1,73 m2)
Assessment of renal function urea | Baseline and follow up (1-31 days after routine surgery if indicated)
  urea (mg/dl)
Assessment of renal function urinary status | Baseline and follow up (1-31 days after routine surgery if indicated)
  standardized urinary status
Assesment of renal function kreatininekinase | Baseline and follow up (1-31 days after routine surgery if indicated)
  kreatininekinase (U/l)

CONTACTS AND LOCATIONS:
Locations (1):
- FAU Erlangen-Nuernberg,, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No